CLINICAL TRIAL: NCT01074333
Title: Prospective, Multicenter, Observational Study on Erbitux® (Cetuximab) in Patients With EGFR-expressing, KRAS Wild-type Metastatic Colorectal Cancer
Brief Title: An Observational Study of Erbitux® in Patients With Metastatic Colorectal Cancer (mCRC) Refractory to Irinotecan-containing Treatment
Status: Terminated | Type: Observational
Why Stopped: This study was terminated due to low recruitment
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR 62202-507
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Colorectal Neoplasm
Keywords: Colorectal cancer; Metastasis; Cetuximab; Erbitux; Epidermal growth factor receptor
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Cetuximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cetuximab — In subjects with mCRC, cetuximab will be used in combination with chemotherapy or as a single agent according to the approved national label as in routine clinical practice. The initial dose of Erbitux is 400 mg/m2 body surface area and the subsequent weekly doses are 250 mg/m2 each administered i.v. via in-line filtration with an infusion pump, gravity drip, or a syringe pump. The recommended infusion period for the initial dose is 120 minutes and for the subsequent weekly doses is 60 minutes with the maximum infusion rate not exceeding 5 ml/min.
  Other Names: Erbitux

SUMMARY:
This is an observational, non-interventional, uncontrolled, multicentric safety study in subjects with epidermal growth factor receptor (EGFR)-expressing, V-Ki-ras2 Kirsten rat sarcoma viral oncogene homolog (KRAS) wild-type mCRC. The study aims to collect safety data related to Erbitux treatment from a total of at least 400 mCRC subjects from about 35 institutions from the start of treatment with Erbitux until progressive disease, Erbitux-related intolerable toxicities, death, or withdrawal of Erbitux treatment (whichever occurs first).

DETAILED DESCRIPTION:
Colorectal cancer is the fourth commonest form of cancer worldwide and remains a leading malignancy both in incidence and mortality. Erbitux is an immunoglobulin G1 monoclonal antibody that specifically blocks ligand binding to the EGFR with high affinity, thereby preventing downstream signal transduction and cellular responses. Erbitux enhances the effects of some common chemotherapy agents and radiotherapy and demonstrates minimal overlapping toxicities with these approaches. Erbitux in combination with other treatment modalities, has also shown efficacy in the treatment of a number of solid tumors, including mCRC, squamous cell carcinoma of the head and neck, and non-small cell lung cancer. Based on several studies conducted in the past, Erbitux has been approved for the treatment of subjects with EGFR-expressing, KRAS wild-type mCRC, as a single agent in subjects who have failed oxaliplatin-and irinotecan-based therapy and who are intolerant to irinotecan or in combination with chemotherapy. The most common Erbitux-related adverse events (AEs) are related to skin, infusion, and hypersensitivity reactions. Other side effects with Erbitux monotherapy include asthenia, dyspnoea, mucositis, nausea, pain, fever and headache.

OBJECTIVES

Primary objective:

* To obtain safety information on the use of Erbitux in subjects with EGFR-expressing, KRAS wild-type mCRC in terms of frequency and severity of AEs

Secondary objective:

* To gather clinical efficacy information of the treatment

The study will primarily collect safety data related to Erbitux treatment along with the clinical efficacy information from the start of treatment with Erbitux until progressive disease, Erbitux related intolerable toxicities, death, or withdrawal of Erbitux treatment whichever occurs first. All subjects will be enrolled in the order to visit the physician after making contract and each subject will be observed for a period of 4 months in average. Erbitux will be prescribed to mCRC subjects according to the approved national label as in routine clinical practice under the supervision of an investigator experienced in the use of antineoplastic medicinal products. Prior to the first infusion, subjects will receive pre-medication with an antihistamine and a corticosteroid. The initial dose of Erbitux is 400 mg/m2 body surface area and the subsequent weekly doses are 250 mg/m2 each administered intravenously (i.v.) via in-line filtration with an infusion pump, gravity drip, or a syringe pump. The recommended infusion period for the initial dose is 120 minutes and for the subsequent weekly doses is 60 minutes with the maximum infusion rate not exceeding 5 ml/min. The observational period of this study is defined as from the first infusion of Erbitux until 28 days after the last infusion of Erbitux in each subject, regardless the reason of discontinuation of Erbitux treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are eligible for Erbitux treatment according to the indication in the national label of Erbitux (i.e. in EGFR expressing, KRAS wild-type metastatic colorectal adenocarcinoma).
* Subjects who have failed oxaliplatin and irinotecan-based therapy and who are intolerant to irinotecan in mCRC.
* Subjects who have signed the informed consent form

Exclusion Criteria:

* Subjects who do not fall under the approved indications according to the national label of Erbitux.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with EGFR-expressing, KRAS wild-type mCRC undergoing treatment with Erbitux in Korea.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2008-09; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Safety and toxicity of Erbitux treatment | 120 minutes and for the subsequent weekly doses is 60 minutes. Before, during and at the end of Erbitux treatment period
  Frequency and severity of all AEs and serious adverse events; Laboratory information (haematology, clinical chemistry, EGFR test and KRAS test).

SECONDARY OUTCOMES:
Clinical efficacy of Erbitux treatment | 120 minutes and for the subsequent weekly doses is 60 minutes From the start of treatment with Erbitux until progressive disease, Erbitux related intolerable toxicities, death, or withdrawal of Erbitux treatment whichever occurs first
  The following data will be collected:
  * Best tumor response with Erbitux treatment
  * Time to progression of tumor with Erbitux treatment
  * Duration of response with Erbitux treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Won Kim, M.D., Ph.D., Principal Investigator — Asan Medical Center, Seoul, Korea, Republic of
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- See also: Related Info — http://globocan.iarc.fr/